CLINICAL TRIAL: NCT03956355
Title: A Phase 3 Efficacy and Safety Study of Tapinarof for the Treatment of Plaque Psoriasis in Adults
Brief Title: Tapinarof for the Treatment of Plaque Psoriasis in Adults (3001)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Organon and Co (Industry)
Collaborators: IQVIA Biotech (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DMVT-505-3001
Record Dates: First submitted 2019-05-16; First posted 2019-05-20 (Actual); Results first posted 2022-10-13 (Actual); Last update posted 2025-06-12 (Actual); Status verified 2022-09

CONDITIONS: Plaque Psoriasis
Keywords: Tapinarof; plaque psoriasis; adult; phase 3; topical; double-blind; efficacy; safety; psoriasis
MeSH Terms: conditions — Psoriasis | interventions — tapinarof

STUDY DESIGN:
Intervention Model Description: Following a 34-day screening period, eligible subjects will be randomized at a 2:1 ratio to receive once daily treatment with tapinarof cream, 1% or vehicle cream.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The Investigator, study center staff, subject, and Sponsor will be blinded to treatment assignment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Tapinarof (DMVT-505) (Experimental): Tapinarof (DMVT-505) Cream Group
  Interventions: Drug: Tapinarof
- Vehicle Cream (Placebo Comparator): Vehicle Cream Group
  Interventions: Drug: Vehicle Cream

INTERVENTIONS:
Drug: Tapinarof — Tapinarof cream, 1%, applied once daily
  Other Names: DMVT-505
  Arms: Tapinarof (DMVT-505)
Drug: Vehicle Cream — Vehicle cream applied once daily
  Arms: Vehicle Cream

SUMMARY:
This is a randomized, double-blind, vehicle-controlled Phase 3 study to evaluate the efficacy and safety of topical tapinarof cream, 1% once daily for the treatment of plaque psoriasis in adults. Approximately 500 adult subjects with plaque psoriasis will be randomized 2:1 to receive either tapinarof cream, 1% or matching vehicle cream once daily for 12 weeks.

DETAILED DESCRIPTION:
This study is a 12-week double-blind, vehicle-controlled treatment study in which subjects will be randomized to receive tapinarof cream, 1% or vehicle cream once daily for 12 weeks. At the end of the 12-week study treatment, qualified subjects completing the study will have the option to enter a separate open-label, long-term safety and efficacy study for an additional 40 weeks of treatment with tapinarof cream, 1%. Subjects who do not enroll in the open-label long-term study will complete a follow-up visit approximately 4 weeks after end of treatment in this study (at Week 16).

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects ages 18 to 75 years with clinical diagnosis of chronic plaque psoriasis and stable disease for at least 6 months prior to the study.
* BSA involvement ≥ 3% and ≤ 20%
* A PGA score of 2 (mild), 3 (moderate) or 4 (severe) at screening and baseline
* Females of child bearing potential and male subjects who are engaging in sexual activity that could lead to pregnancy agree to follow the specified contraceptive guidance throughout the study, including screening, during the treatment period, and for at least 4 weeks after the last exposure to study treatment
* Capable of giving written informed consent

Exclusion Criteria:

* Psoriasis other than plaque variant
* Any sign of infection of any of the psoriatic lesions
* Concurrent conditions or history of other diseases:
* Immunocompromised at Screening
* Chronic or acute infection requiring treatment with systemic antibiotics, antivirals, antiparasitics, antiprotozoals, or antifungals within 4 weeks prior to the Baseline visit
* Acute active bacterial, fungal, or viral (herpes simplex, herpes zoster, chicken pox) skin infection within 1 week prior to the Baseline visit
* Significant dermatologic or inflammatory condition other than plaque psoriasis that, in the Investigator's opinion, would make it difficult to interpret data or assessments during the study
* Alanine aminotransferase (ALT) or aspartate aminotransferase (AST) ≥ 1.5x the upper limit of normal (ULN)
* Total bilirubin > 1.5 x ULN; total bilirubin > ULN and ≤ 1.5 x ULN is acceptable if bilirubin is fractionated and direct bilirubin < 35%
* Corrected QT interval > 475
* Current or chronic history of liver disease, known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones), presence of hepatitis B surface antigen (HBsAg), or positive hepatitis C antibody test result, or a positive anti-hepatitis B core antigen (anti-HBc) result
* Ultraviolet (UV) light therapy or prolonged exposure to natural or artificial sources of UV radiation within 4 weeks prior to the Baseline visit and/or plans to have such exposures during the study which could potentially impact the subject's psoriasis
* Use of any prohibited medication within the indicated period before the first dose of study drug
* Within a minimum of 5 half-lives for biologic agents:
* Within 4 weeks for systemic immunosuppressive or immunomodulating agents, fumaric acid derivatives, vitamin D3 and analogs, retinoids, psoralens, corticosteroids, adrenocorticotropic hormone analogs, and tazarotene
* 2 weeks for immunizations with a live viral component; drugs known to possibly worsen psoriasis, unless on a stable dose for > 12 weeks
* With the exception of non-medicated emollients, 2 weeks for topical treatments including corticosteroids, immunomodulators, anthralin (dithranol), vitamin D derivatives or coal tar.
* Pregnant females or lactating females
* History of sensitivity to the study drugs, or components thereof or a history of drug or other allergy that, in the opinion of the Investigator or Medical Monitor, contraindicates the subject's participation in the study
* The subject has received an investigational product within 30 days, 5 half-lives, or twice the duration of the biological effect of the study drug (whichever is longer) prior to first dose of study drug
* Current or a history of cancer within 5 years except for fully excised skin basal cell carcinoma, squamous cell carcinoma or carcinoma in situ of the cervix
* Subjects with active infection that required oral, intramuscular, or intravenous administration of antibiotics, antifungal or antiviral agents within 7 days of Baseline/Day 1
* Previous known participation in a clinical study with tapinarof
* Evidence of significant hepatic, renal, respiratory, endocrine, hematologic, neurologic, psychiatric, or cardiovascular (CV) system abnormalities or laboratory abnormality that will affect the health of the subject or interfere with interpretation of the results

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 510 (Actual)
Dates: Start 2019-05-21 (Actual); Primary Completion 2020-05-26 (Actual); Study Completion 2020-05-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Victoria Butners, Study Director — Dermavant Sciences GmbH
Locations (52):
- United States (43):
  - Dermavant Investigative Site, Birmingham, Alabama
  - Dermavant Investigative Site, Phoenix, Arizona
  - Dermavant Investigative Site, Hot Springs, Arkansas
  - Dermavant Investigative Site, Rogers, Arkansas
  - Dermavant Investigative Site, Anaheim Hills, California
  - Dermavant Investigative Site, Fresno, California
  - Dermavant Investigative Site, Los Angeles, California
  - Dermavant Investigative Site, Northridge, California
  - Dermavant Investigative Site, San Diego, California
  - Dermavant Investigative Site, Santa Ana, California
  - Dermavant Investigative Site, Cromwell, Connecticut
  - Dermavant Investigative Site, Boca Raton, Florida
  - Dermavant Investigative Site, Brandon, Florida
  - Dermavant Investigative Site, Hialeah, Florida
  - Dermavant Investigative Site, Miramar, Florida
  - Dermavant Investigative Site, Marietta, Georgia
  - Dermavant Investigative Site, Evansville, Indiana
  - Dermavant Investigative Site, Indianapolis, Indiana
  - Dermavant Investigative Site, New Albany, Indiana
  - Dermavant Investigative Site, Louisville, Kentucky
  - Dermavant Investigative Site, Owensboro, Kentucky
  - Dermavant Investigative Site, Baton Rouge, Louisiana
  - Dermavant Investigative Site, New Orleans, Louisiana
  - Dermavant Investigative Site, Boston, Massachusetts
  - Dermavant Investigative Site, Clarkston, Michigan
  - Dermavant Investigative Site, Warren, Michigan
  - Dermavant Investigative Site, Saint Joseph, Missouri
  - Dermavant Investigative Site, Verona, New Jersey
  - Dermavant Investigative Site, Kew Gardens, New York
  - Dermavant Investigative Site, New York, New York
  - Dermavant Investigative Site, Rochester, New York
  - Dermavant Investigative Site, Cary, North Carolina
  - Dermavant Investigative Site, High Point, North Carolina
  - Dermavant Investigative Site, Norman, Oklahoma
  - Dermavant Investigative Site, Portland, Oregon
  - Dermavant Investigative Site, Pittsburgh, Pennsylvania
  - Dermavant Investigative Site, Johnston, Rhode Island
  - Dermavant Investigative Site, Arlington, Texas
  - Dermavant Investigative Site, College Station, Texas
  - Dermavant Investigative Site, Dripping Springs, Texas
  - Dermavant Investigative Site, Houston, Texas
  - Dermavant Investigative Site, San Antonio, Texas
  - Dermavant Investigative Site, West Jordan, Utah
- Canada (9):
  - Dermavant Investigative Site, Saint Johns, Newfoundland and Labrador
  - Dermavant Investigative Site, Ajax, Ontario
  - Dermavant Investigative Site, Coburg, Ontario
  - Dermavant Investigative Site, North Bay, Ontario
  - Dermavant Investigative Site, Richmond Hill, Ontario
  - Dermavant Investigative Site, Toronto, Ontario
  - Dermavant Investigative Site, Waterloo, Ontario
  - Dermavant Investigative Site, Windsor, Ontario
  - Dermavant Investigative Site, Montreal, Quebec

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Lebwohl MG, Stein Gold L, Strober B, Papp KA, Armstrong AW, Bagel J, Kircik L, Ehst B, Hong HC, Soung J, Fromowitz J, Guenthner S, Piscitelli SC, Rubenstein DS, Brown PM, Tallman AM, Bissonnette R. Phase 3 Trials of Tapinarof Cream for Plaque Psoriasis. N Engl J Med. 2021 Dec 9;385(24):2219-2229. doi: 10.1056/NEJMoa2103629. PMID 34879448
- [Derived] Gold LS, Bruno MJ, Lewitt GM, Hebert AA. Characteristics and management of follicular events and contact dermatitis in patients using tapinarof cream for the treatment of atopic dermatitis or plaque psoriasis. J Dermatolog Treat. 2025 Dec;36(1):2517388. doi: 10.1080/09546634.2025.2517388. Epub 2025 Jul 2. PMID 40600584
- [Derived] Kircik L, Zirwas M, Kwatra SG, Lewitt GM, Glover H, Chao T, Brown PM, Rubenstein DS, Tallman AM. Rapid Improvements in Itch with Tapinarof Cream 1% Once Daily in Two Phase 3 Trials in Adults with Mild to Severe Plaque Psoriasis. Dermatol Ther (Heidelb). 2024 Jan;14(1):201-211. doi: 10.1007/s13555-023-01068-x. Epub 2023 Dec 21. PMID 38123875
- [Derived] Desai SR, Stein Gold L, Cameron MC, Golant A, Lewitt GM, Bruno MJ, Martin G, Brown PM, Rubenstein DS, Butners V, Tallman AM. Tapinarof Cream 1% Once Daily for the Treatment of Plaque Psoriasis: Case Photography of Clinical Outcomes from Three Phase 3 Trials. Dermatol Ther (Heidelb). 2023 Oct;13(10):2443-2460. doi: 10.1007/s13555-023-01008-9. Epub 2023 Sep 11. PMID 37697121

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Tapinarof (DMVT-505) | Vehicle Cream
Started | 340 | 170
Completed | 269 | 130
Not Completed | 71 | 40

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Tapinarof (DMVT-505) | Vehicle Cream | Total
Number analyzed (Participants) | 340 | 170 | 510
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.8 (13.68) | 49.1 (13.25) | 49.6 (13.53)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 127 | 84 | 211
  Male | 213 | 86 | 299
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 53 | 34 | 87
  Not Hispanic or Latino | 284 | 135 | 419
  Unknown or Not Reported | 3 | 1 | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 21 | 4 | 25
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 18 | 11 | 29
  White | 286 | 146 | 432
  More than one race | 10 | 7 | 17
  Unknown or Not Reported | 4 | 2 | 6
Physician Global Assessment [Count of Participants; unit: Participants] — The PGA is a clinical tool for assessing the current state/severity of a subject's psoriasis at a given timepoint. A static 5-point scale is used to grade lesions on the clinical characteristics of erythema, scaling, and plaque thickness/elevation. The PGA ranges from 0 to 4, and is calculated as Clear (0), Almost clear (1), Mild (2), Moderate (3), and Severe (4). Higher PGA scores represent more severe disease.
  Participants
    0 - clear | 0 | 0 | 0
    1 - almost clear | 0 | 0 | 0
    2 - mild | 39 | 21 | 60
    3 - moderate | 271 | 133 | 404
    4 - severe | 30 | 16 | 46
Psoriasis Area and Severity Index [Mean (Standard Deviation); unit: units on a scale] — The Psoriasis Area and Severity Index (PASI) scoring system combines lesion severity and extent of affected area into 1 score: 0 (no disease) to 72 (maximal disease). 4 areas (head, arms, trunk, and legs) are each assessed for 3 signs: erythema (redness), induration (plaque thickness), and scale using a 5-point scale, where 0=none, 1=slight, 2=mild, 3=moderate, 4=severe and percent of skin involved using a 6-point scale were 6 is worse. Scores are multiplied by a weighted factor for each region; the sum of these scores gives the overall PASI score. Higher scores indicate more severe disease.
  units on a scale | 8.71 (3.979) | 9.19 (4.395) | 8.87 (4.124)
Percent Body Surface Area [Mean (Standard Deviation); unit: Percent] — The handprint method was used to assess BSA with psoriasis, where the full palmar hand of the participant represented approximately 1% of the total BSA. Body regions are assigned specific number of handprints with percentage [Head and neck = 10% (10 handprints), upper extremities = 20% (20 handprints), Trunk (including axillae and groin) = 30% (30 handprints), lower extremities (including buttocks) = 40% (40 handprints)]. Estimates of the % involvement in each body region will be multiplied by the fraction of total body area to obtain the total %BSA involved by region and overall.
  Percent | 7.8 (4.64) | 8.2 (5.06) | 7.9 (4.78)

OUTCOME MEASURES:

1. Primary Outcome: Percent of Subjects Who Achieve a Physician Global Assessment (PGA) Score of Clear (0) or Almost Clear (1) With a Minimum 2-grade Improvement From Baseline at Week 12. Analyses Were Done Using Multiple Imputation
Description: The PGA is a clinical tool for assessing the current state/severity of a subject's psoriasis at a given timepoint. A static 5-point scale is used to grade lesions on the clinical characteristics of erythema, scaling, and plaque thickness/elevation. The PGA ranges from 0 to 4, and is calculated as Clear (0), Almost clear (1), Mild (2), Moderate (3), and Severe (4). Higher PGA scores represent more severe disease. Analyses were done using multiple imputation.
Time Frame: Baseline to Week 12
Measure: Mean (Standard Error); unit: percentage of subjects
Arm/Group | Tapinarof (DMVT-505) | Vehicle Cream
Number analyzed (Participants) | 340 | 170
percentage of subjects | 35.4 (2.75) | 6.0 (2.08)
Statistical Analysis 1: Comparison: Tapinarof (DMVT-505) vs Vehicle Cream; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel; Risk Ratio (RR) = 5.78

2. Secondary Outcome: Percent of Subjects With ≥ 75% Improvement in Psoriasis Area and Severity Index (PASI) From Baseline at Week 12. Analyses Were Done Using Multiple Imputation.
Description: The Psoriasis Area and Severity Index (PASI) scoring system combines the assessment of lesion severity and extent of affected area into a single score: 0 (no disease) to 72 (maximal disease). The body is divided into 4 areas for scoring (head, arms, trunk, and legs). Each area is assessed for 3 signs: erythema (redness), induration (plaque thickness), and scale. The severity of each sign in each body area is assessed and scored independently using a 5-point scale, where 0=none, 1=slight, 2=mild, 3=moderate, 4=severe. Each area is also assessed for percent of skin involved: 0 = (0%), 1 = (1-<10%), 2 = (10-<30%), 3 = (30-<50%), 4 = (50 -<70%), 5 = (70-<90%), 6 = (90-100%). The individual scores are multiplied by a weighted factor for each body region; the sum of these scores gives the overall PASI score. Higher scores indicate more severe disease. PASI is a static assessment made without reference to previous scores. Analyses were done using multiple imputation.
Time Frame: Baseline to Week 12
Measure: Mean (Standard Error); unit: percentage of subjects
Arm/Group | Tapinarof (DMVT-505) | Vehicle Cream
Number analyzed (Participants) | 340 | 170
percentage of subjects | 36.1 (2.73) | 10.2 (2.43)
Statistical Analysis 1: Comparison: Tapinarof (DMVT-505) vs Vehicle Cream; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel; Risk Ratio (RR) = 2.76

3. Secondary Outcome: Percent of Subjects With a PGA Score of 0 or 1 at Week 12. Analyses Were Done Using Multiple Imputation.
Description: as for outcome 1
Time Frame: Baseline to Week 12
Measure: Mean (Standard Error); unit: percentage of subjects
Arm/Group | Tapinarof (DMVT-505) | Vehicle Cream
Number analyzed (Participants) | 340 | 170
percentage of subjects | 37.8 (2.79) | 9.9 (2.51)
Statistical Analysis 1: Comparison: Tapinarof (DMVT-505) vs Vehicle Cream; Test type: Superiority; p = 0.0001, Cochran-Mantel-Haenszel; Risk Ratio (RR) = 2.68

4. Secondary Outcome: Mean Change in Percent of Total Body Surface Area (%BSA) Affected From Baseline to Week 12
Description: Assessment of BSA with psoriasis was estimated by means of the handprint method, where the full palmar hand of the participant (fully extended palm, fingers and thumb together) represented approximately 1% of the total BSA. Body regions are assigned specific number of handprints with percentage [Head and neck = 10% (10 handprints), upper extremities = 20% (20 handprints), Trunk (including axillae and groin) = 30% (30 handprints), lower extremities (including buttocks) = 40% (40 handprints)]. Estimates of the % involvement in each body region will be multiplied by the fraction of total body area to obtain the total %BSA involved by region and overall.
Time Frame: Baseline to Week 12
Measure: Least Squares Mean (Standard Error); unit: Mean change from Baseline
Arm/Group | Tapinarof (DMVT-505) | Vehicle Cream
Number analyzed (Participants) | 340 | 170
Mean change from Baseline | -3.50 (0.471) | -0.22 (0.579)
Statistical Analysis 1: Comparison: Tapinarof (DMVT-505) vs Vehicle Cream; Test type: Superiority; p < 0.0001, ANCOVA; Least squares mean difference = -3.28

5. Secondary Outcome: Percent of Subjects With ≥90% Improvement in PASI Score From Baseline to Week 12. Analyses Were Done Using Multiple Imputation.
Description: as for outcome 2
Time Frame: Baseline to Week 12
Measure: Mean (Standard Error); unit: percentage of subjects
Arm/Group | Tapinarof (DMVT-505) | Vehicle Cream
Number analyzed (Participants) | 340 | 170
percentage of subjects | 18.8 (2.18) | 1.6 (1.05)
Statistical Analysis 1: Comparison: Tapinarof (DMVT-505) vs Vehicle Cream; Test type: Superiority; p = 0.0005, Cochran-Mantel-Haenszel; Risk Ratio (RR) = 8.54

ADVERSE EVENTS:
Time Frame: Subject duration: 12 weeks of treatment and 4 week follow-up for subjects not enrolled in the long-term extension study (DMVT-505-3003)
Groups:
- Tapinarof (DMVT-505): Tapinarof (DMVT-505) Cream Group
  Tapinarof: Tapinarof cream, 1%, applied once daily.
  All SAEs were deemed unrelated to treatment with tapinarof cream, 1%.
- Vehicle Cream: Vehicle Cream Group
  Vehicle Cream: Vehicle cream applied once daily.
  All SAEs were deemed unrelated to treatment with tapinarof cream, 1%.
Arm/Group | Tapinarof (DMVT-505) | Vehicle Cream
All-Cause Mortality (participants affected / at risk) | 0/340 | 0/170
Serious Adverse Events (participants affected / at risk) | 9/340 | 0/170
Other Adverse Events (participants affected / at risk) | 131/340 | 27/170
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Tapinarof (DMVT-505) (N=340) | Vehicle Cream (N=170)
Cardiac failure congestive (Cardiac disorders) | 1 | 0
Coronary artery disease (Cardiac disorders) | 1 | 0
Pericardial effusion (Cardiac disorders) | 1 | 0
Oesophageal obstruction (Gastrointestinal disorders) | 1 | 0
Pancreatitis acute (Gastrointestinal disorders) | 1 | 0
Cellulitis (Infections and infestations) | 1 | 0
Stab wound (Injury, poisoning and procedural complications) | 1 | 0
Laryngospasm (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Aortic arteriosclerosis (Vascular disorders) | 1 | 0
Hypertensive crisis (Vascular disorders) | 1 | 0
Hypertensive urgency (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Tapinarof (DMVT-505) (N=340) | Vehicle Cream (N=170)
abdominal pain (Gastrointestinal disorders) | 4 | 0
Folliculitis (Infections and infestations) | 79 | 2
Nasopharyngitis (Infections and infestations) | 25 | 10
Upper respiratory tract infection (Infections and infestations) | 5 | 4
Viral upper respiratory tract infection (Infections and infestations) | 7 | 2
Influenza (Infections and infestations) | 5 | 0
Cystitis (Infections and infestations) | 0 | 2
Ligament sprain (Injury, poisoning and procedural complications) | 1 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 4 | 2
Headache (Nervous system disorders) | 10 | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 4 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Dermatitis contact (Skin and subcutaneous tissue disorders) | 15 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 8 | 0
Rash (Skin and subcutaneous tissue disorders) | 4 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2019-08-08): https://cdn.clinicaltrials.gov/large-docs/55/NCT03956355/Prot_000.pdf
  • Statistical Analysis Plan (2020-05-04): https://cdn.clinicaltrials.gov/large-docs/55/NCT03956355/SAP_001.pdf